CLINICAL TRIAL: NCT03707678
Title: A Multicentre, Randomised, Placebo-controlled, Double-blind (Sponsor Open), Parallel-group, 8-week Treatment Study Investigating the Efficacy and Safety of Intra-nasal GSK2245035 in Adults With Allergic Asthma Treated With Inhaled Corticosteroids (ICS)
Brief Title: A Safety and Efficacy Study of Intranasal GSK2245035 in Adults With Allergic Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: After careful review of new data on GSK2245035, GlaxoSmithKline has decided to cancel this study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207542
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: GSK2245035; Allergic asthma; Inhaled corticosteroids; Toll-like receptors
MeSH Terms: conditions — Asthma | interventions — GSK2245035; Albuterol

STUDY DESIGN:
Intervention Model Description: This will be a parallel-group study. Subjects will be randomized in 1:1 ratio to receive GSK2245035 or placebo once weekly for 8 weeks.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study where the investigators and subjects will be blinded and sponsor remains unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects receiving GSK2245035 (Experimental): Eligible subjects will be administered 20 nanograms (ng) of GSK2245035 nasal spray solution using a metered Valois VP7 pump (1 spray=10 ng per actuation per nostril) once weekly for 8 weeks. Subjects will also receive tapering doses of FP-DPI 100-500 mcg twice daily during the treatment period. Albuterol/Salbutamol metered dose inhaler (MDI) will be given for symptom relief from screening to the end of the study.
  Interventions: Drug: GSK2245035; Drug: FP-DPI; Drug: Albuterol/Salbutamol; Other: eDairy; Other: ACQ-6
- Subjects receiving placebo (Placebo Comparator): Eligible subjects will be administered placebo nasal spray solution using a metered Valois VP7 pump (1 spray per actuation per nostril) once weekly for 8 weeks. Subjects will also receive tapering doses of FP-DPI 100-500 mcg twice daily during the treatment period. Albuterol/Salbutamol MDI will be given for symptom relief from screening to the end of the study.
  Interventions: Drug: Placebo; Drug: FP-DPI; Drug: Albuterol/Salbutamol; Other: eDairy; Other: ACQ-6

INTERVENTIONS:
Drug: GSK2245035 — GSK2245035 will be administered weekly once as a nasal spray solution with dosing strength of 10 ng per actuation. GSK2245035 will be available as a saline formulation, preserved with benzalkonium chloride and disodium edetate in an amber glass bottle fitted with a screw-fit atomizing pump.
  Arms: Subjects receiving GSK2245035
Drug: Placebo — Placebo will be administered weekly once as a nasal spray solution. Placebo will be available as a saline formulation, preserved with benzalkonium chloride and disodium edetate in an amber glass bottle fitted with a screw-fit atomizing pump.
  Arms: Subjects receiving placebo
Drug: FP-DPI — FP will be administered using Diskus inhaler with dosing strengths of 500, 250, 100, 50 µg twice daily per actuation.
Drug: Albuterol/Salbutamol — Albuterol/Salbutamol MDI will be administered for symptom relief from screening to the end of the study.
Other: eDairy — Subjects will record all the alerts indicative of worsening of asthma in eDairy.
Other: ACQ-6 — ACQ-6 will include six questions which enquire about the frequency and/or severity of symptoms. The response options for all these questions consist of a zero (no impairment/limitation) to six (total impairment/limitation) scale.

SUMMARY:
GSK2245035 belongs to a novel class of agonist drugs targeted at toll like receptors (TLR). T-helper cell 2 (Th2) driven inflammation is a key patho-physiological mechanism in allergic asthma. The clinical manifestations and inflammatory pathways of allergic asthma are sensitive to corticosteroid therapy. However, GSK2245035 reduces Th2-driven airway inflammation and thereby controls asthma symptoms. This study aims to determine whether intranasal GSK2245035 maintains biological and clinical control of allergic asthma using 'tapering of ICS' study design. This study will assess the efficacy and safety of GSK2245035 in subjects with allergic asthma treated with ICS. This will be a randomised, double-blind (sponsor open), placebo-controlled, parallel group, 8-week study treatment period. The study will consist of a screening period of up to approximately 5 weeks, blinded treatment period of 8 weeks, followed by a follow-up period of 7 weeks. A total of 60 subjects will be included in this study and duration of time for each subject will therefore be 141 days including screening and study ICS dose adjustment period. Diskus® is a registered trademark of GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Physician confirmed diagnosis of asthma for at least 6 months prior to screening.
* Asthma therapy with inhaled corticosteroids (fluticasone propionate dry powder inhaler [FP-DPI] >=100 micrograms (mcg), or equivalent, total daily dose) >=3 months (at time screening visit 1 [SV1]).
* Body weight >= 45 kilograms (kg).
* Male or female of non-reproductive potential. A male subject must agree to use a highly effective contraception during the treatment period and at least from the time of first dose of study medication until the final follow-up visit and refrain from donating sperm during this period. A female subject is eligible to participate if she is not a woman of childbearing potential (WOCBP).
* Capable of giving signed informed consent.

Exclusion Criteria:

* Current smokers or former smokers with a smoking history >=10 pack years.
* Clinically significant abnormal laboratory result (Chemistry, Hematology and Urinalysis) at SV1.
* Alanine transaminase (ALT) >2xupper limit of normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Clinically significant and abnormal electrocardiogram (ECG) at screening visit 1.
* Heart rate corrected QT interval (QTc) > 450 milliseconds (msec) or QTc > 480 msec in subject with Bundle Branch Block.
* Subjects with a diagnosis of malignancy or in the process of investigation for a malignancy.
* Subjects on oral corticosteroid therapy.
* Subjects who have received treatment with allergen immunotherapy (in the last 2 years), anti-immunoglobulin E (IgE) or anti interleukin 5 (IL5) or anti IL13 antibodies or immunosuppressive agents (example given [e.g.] methotrexate, azothioprine, cyclosporine) within the past 6 months.
* A pre-bronchodilator forced expiratory volume in 1 second (FEV1) < 50 percent predicted of normal value.
* Occupational asthma due to low molecular weight chemicals.
* Asthma exacerbation requiring treatment with systemic corticosteroids or hospitalization within 3 months prior to screening.
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 10 years.
* Evidence of concurrent respiratory diseases such as pneumonia, tuberculosis, pneumothorax, atelectasis, pulmonary fibrotic disease, allergic bronchopulmonary aspergillosis, cystic fibrosis, bronchopulmonary dysplasia, or other respiratory abnormalities other than asthma.
* Respiratory tract infection that is not resolved within 2 weeks prior to screening.
* Other conditions that could lead to elevated eosinophils such as hypereosinophilic syndromes. Subjects with a known, pre-existing parasitic infestation within 6 months prior to screening.
* A current or past diagnosis of an autoimmune disorder such as systemic lupus erythematosus (SLE).
* Other concurrent diseases/abnormalities: A subject must not have any clinically significant uncontrolled condition, or disease state, that, in the opinion of the investigator, would put the safety of the subject at risk through study participation. E.g. Addison's disease hypertension 1 (uncontrolled) aortic aneurysm (clinically significant), peptic ulcer (recent or poorly controlled), Cushing's disease, renal disease, diabetes mellitus (uncontrolled), stroke within 3 months of screening visit 1, thyroid disorder (uncontrolled), hepatic disease tuberculosis (current or untreated).
* History of sensitivity to any of the study medications, including Albuterol/Salbutamol or Albuterol components there of or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of hypersensitivity to investigational medicinal product (IMP) or to drugs of similar chemical class (TLR agonists).
* The subject has received an investigational medicinal product within 30 days or, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer). Use of a biologic (e.g. monoclonal antibodies) agent for the treatment of asthma in the past 6 months.
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.
* Presence of hepatitis B surface antigen (HbsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Known positive for Human Immunodeficiency Virus (HIV) antibody.
* Donation or loss of 400 milliliters (mL) or more of blood within 8 weeks prior to initial dosing, or longer if required by local regulation or hemoglobin levels below normal range at screening or where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 units for males and females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* A history of substance abuse including alcohol.
* Subjects at risk of non-compliance, or unable to comply with the study procedures.
* Subjects who are unable to follow study instructions such as visit schedule, dosing directions, study electronic diary (eDiary) completion, or use of a standard metered dose inhaler. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-21 (Estimated); Primary Completion 2019-12-23 (Estimated); Study Completion 2019-12-23 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in fractional exhaled breath nitric oxide (FeNO) level | Baseline and up to Week 9
  FeNO level will be measured to determine efficacy of GSK2245035 in reducing asthma (airway) inflammation. The measurements will be performed using a handheld electronic device. 'Primary Endpoint Visit' (PEPV) will be 1-week post 8th dose. Subjects withdrawn from the study before PEPV because of protocol defined asthma worsening will attend a 'treatment withdrawal visit'.

SECONDARY OUTCOMES:
Number of subjects experiencing worsening of asthma from Baseline to PEPV | Baseline and up to Week 9
  Asthma worsening is defined as one or more of the following: an increase in asthma control questionnaire 6 (ACQ-6) >0.5 from Baseline; a daily asthma symptom score of >=4 for 2 consecutive days; nocturnal awaking(s) due to asthma requiring short-acting beta agonist (SABA) use on 2 consecutive nights; an increase from Baseline of >=4 puffs per day of rescue medication use on 2 consecutive days; >=20 percent reduction in morning peak expiratory flow (PEF) from Baseline and >=20 percent reduction in evening PEF from Baseline for 2 consecutive days; visit to emergency room / department, hospitalization or oral corticosteroid therapy for severe asthma exacerbation.
Time for FeNO to increase by 10 parts per billion (ppb) | Up to Week 15
  Increase in FeNO by 10 ppb will be calculated from first dose of GSK2245035 or placebo up to the 'study completion visit'.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com